CLINICAL TRIAL: NCT01458977
Title: Prospective, Randomised, Crossover, Double-Blind, Placebo-Controlled Trial To Assess The Lipid-Lowering Effect Of Adding Tenofovir/Emtricitabine Co-Formulation Vs Placebo To Hiv-1-Infected Subjects With Dyslipidemia And Sustained Viral Load Suppression Under Monotherapy With Ritonavir-Boosted Protease Inhibitors
Brief Title: Trial To Assess The Lipid-Lowering Effect Of Adding Tenofovir/Emtricitabine Co-Formulation Vs Placebo To Hiv-1-Infected Subjects With Dyslipidemia And Sustained Viral Load Suppression Under Monotherapy With Ritonavir-Boosted Protease Inhibitors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TULIP
Record Dates: First submitted 2011-10-21; First posted 2011-10-25 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: HIV; Dyslipidemia
Keywords: Lípid-lowering effect; Tenofovir; Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TDF/FTC (3 months) + Placebo (6 months) (Experimental): TDF/FTC (3 months) + Placebo (6 months)
  Interventions: Drug: Truvada® (300 mg tenofovir disoproxil fumarato/200 mg emtricitabine)
- Placebo (3 months) + TDF/FTC (3 months) + Placebo (3 months) (Placebo Comparator): Placebo (3 months) + TDF/FTC (3 months) + Placebo (3 months)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Truvada® (300 mg tenofovir disoproxil fumarato/200 mg emtricitabine) — TDF/FTC 300/200mg daily during 3 months + Placebo during 6 months
  Other Names: N/H
  Arms: TDF/FTC (3 months) + Placebo (6 months)
Drug: Placebo — Placebo during 3 months + TDF/FTC 300/200mg daily during 3 months + Placebo during 3 months
  Other Names: N/H
  Arms: Placebo (3 months) + TDF/FTC (3 months) + Placebo (3 months)

SUMMARY:
This is a phase IV, multicenter, prospective, randomised, crossover, double blind, placebo-controlled and proof of concept clinical trial.

All subjects fulfilling inclusion criteria will be randomised to add either TDF/FTC co-formulation (group A) or placebo (Group B) to their current PI/r regimen, i.e.: DRV/r 800/100 mg QD or LPV/r 400/100 BID. This will be followed by a crossover addition of TDF/FTC co-formulation or placebo.

Randomization will be centralised in the CRO FLS-Research Support and will be stratified by DRV/r or LPV/r intake at baseline to ensure equal distribution in both arms. TDF/FTC co-formulation or Placebo will be provided in a double-blinded fashion, i.e.: neither the treating physician nor the patient will know whether the patient is receiving TDF/FTC or placebo.

All subjects will receive dietary counselling to promote lipid-lowering diet provided by a specialised dietician throughout the study.

The expected duration of the study for each participant will be 36 weeks. There will be 6 visits: screening, baseline and weeks 4, 12, 24 and 36.

DETAILED DESCRIPTION:
This is a phase IV, multicenter,, prospective, randomised, crossover, double blind, placebo-controlled and proof of concept clinical trial. The trial was conducted in a total sample of 60 patients (30 patients per group), which assures adequate power to detect differences. This study is adequate to demonstrate the lipid-lowering effect of TDF/FTC co-formulation addition in patients with dyslipidemia and stable monotherapy antiretroviral treatment.

All subjects fulfilling inclusion criteria will be randomised to add either TDF/FTC co-formulation (group A) or placebo (Group B) to their current PI/r regimen, i.e.: DRV/r 800/100 mg QD or LPV/r 400/100 BID. This will be followed by a crossover addition of TDF/FTC co-formulation or placebo.

In Group A the expected changes in cholesterol values, regarding baseline, can be observed 3 months after TDF/FTC addition. After this, a period of 3 months with placebo will act as a washout period, allowing establishing comparisons intra-patient. Finally, another period of 3 months with placebo will permit to establish comparisons with the first 3-month TDF/FTC intervention. In Group B, subjects will follow a 3-month placebo period, later a 3-month TDF/FTC intervention and finally a placebo period that will act as a wash-out.

Randomization will be centralised in the CRO FLS-Research Support and will be stratified by DRV/r or LPV/r intake at baseline to ensure equal distribution in both arms. TDF/FTC co-formulation or Placebo will be provided in a double-blinded fashion, i.e.: neither the treating physician nor the patient will know whether the patient is receiving TDF/FTC or placebo.

All subjects will receive dietary counselling to promote lipid-lowering diet provided by a specialised dietician throughout the study.

The expected duration of the study for each participant will be 36 weeks. There will be 6 visits: screening, baseline and weeks 4, 12, 24 and 36.

The date for the inclusion of the first patient was November 2011 and the end of the last patient follow-up has been in February 2014. The enrolment period has been 18 months. The final study report will be submitted before November 2014.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Chronic HIV-1 infection
3. Antiretroviral treatment with either DRV/r (800/100 mg QD) or LPV/r (400/100 mg BID) monotherapy during at least 6 months prior to screening.
4. Fasting total cholesterol or LDL-cholesterol levels ≥ 200 and ≥130 mg/dL respectively, in the previous two consecutive tests obtained at least 4 weeks apart before screening.
5. Calculated creatinine clearance ≥ 60 mL/min, according to the Cockcroft-Gault formula.
6. Undetectable plasma HIV-1 RNA levels (< 50 copies/mL) during at least 6 months prior to screening.
7. Adequate treatment adherence.
8. Absence of TDF or FTC resistances.
9. Written informed consent to participate into the study.

Exclusion Criteria:

1. Acute infections or uncontrolled chronic infection in the 2 months previous to the inclusion or physical examination that, in the investigator's opinion, would compromise the patient's safety or outcome of the study
2. Lactating, pregnancy or fertile women willing to be pregnant.
3. Concomitant use of any drug with potential drug-drug interaction with DRV/r, LPV/r or TDF/FTC co-formulation at study entry.
4. Concomitant use of any lipid-lowering drugs at study entry.
5. Prior documented intolerance or hypersensitivity to TDF, FTC, LPV/r or DRV/r.
6. Therapies including interferon, interleukin-2, cytotoxic chemotherapy or immunosuppressors at study entry.
7. Acute or chronic renal documented pathologies.
8. Documented resistance to any of the study drugs (either genotypic or phenotypic)
9. Life expectancy less or equal to 1 year.
10. Current alcohol or substance use judged by the investigator to potentially interfere with subject study compliance.
11. Subjects currently taking part in any other clinical trial using an investigational product, with the exception of studies where the treatment studied have stopped for more than 12 weeks.
12. Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the subject unsuitable for the study or unable to comply with the dosing requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Total fasting cholesterol | Baseline, week 4, 12, 24 and 36
LDL-cholesterol | Baseline, week 4, 12, 24 and 36

SECONDARY OUTCOMES:
CD4 cell count | Baseline, week 4, 12, 24 and 36
Changes in liver enzymes | Baseline, week 4, 12, 24 and 36
Changes in phosphate | Baseline, week 4, 12, 24 and 36
Changes in creatinine | Baseline, week 4, 12, 24 and 36
Changes in glomerular filtration rate | Baseline, week 4, 12, 24 and 36
Changes in HDL cholesterol | Baseline, week 4, 12, 24 and 36
Changes in triglycerides | Baseline, week 4, 12, 24 and 36
Adverse events | Baseline, week 4, 12, 24 and 36
Resistance mutations | Baseline, week 4, 12, 24 and 36
lipid-lowering drugs | Baseline, week 4, 12, 24 and 36

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Germans Trias i Pujol Hospital, Badalona, Barcelona
  - Hospital Valle Hebrón, Barcelona, Barcelona
  - Hospital de Bellvitge, L'Hospitalet de Llobregat, Barcelona

REFERENCES:
- [Derived] Santos JR, Saumoy M, Curran A, Bravo I, Llibre JM, Navarro J, Estany C, Podzamczer D, Ribera E, Negredo E, Clotet B, Paredes R; Tenofovir/emtricitabine inflUence on LIPid metabolism (TULIP) Study Group. The lipid-lowering effect of tenofovir/emtricitabine: a randomized, crossover, double-blind, placebo-controlled trial. Clin Infect Dis. 2015 Aug 1;61(3):403-8. doi: 10.1093/cid/civ296. Epub 2015 Apr 13. PMID 25870325